CLINICAL TRIAL: NCT02789072
Title: Effects of Microgravity on Central Aortic Pressure During Parabolic Flights
Acronym: CapFlight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Novespace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A01259-40
Record Dates: First submitted 2016-04-21; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microgravity (Other): effect of microgravity on central aortic blood pressure.
  Interventions: Other: central aortic pressure (measured in mmHg).

INTERVENTIONS:
Other: central aortic pressure (measured in mmHg). — Blood pressure will only be measured during the 0g (microgravity) phase. Seven 5 ml blood sample will be drawn in the aircraft: before the first parabola (1) and after each block of 5 parabola (6).
  On ground after flight, a 9th 5 ml blood sample will be drawn and then the mobil-o-graph, the SOMNOtouch NIBP and the intravenous cannula will be removed.

SUMMARY:
Cardiovascular events remain the main cause of death of the industrialized world (Global status report on noncommunicable diseases 2010. Geneva, World Health Organization, 2011). Arterial hypertension, hyperlipoproteinemia, smoking, diabetes and family history represent the main cardiovascular risk factors. Arteriosclerosis leads to coronary heart disease, cerebrovascular insufficiency and peripheral vascular diseases that reflect in myocardial infarction and stroke.

The main objective of this experiment is to investigate the differential effect of microgravity on central aortic blood pressure.

The main criterion is the central aortic pressure (measured in mmHg). The hypothesis is that microgravity leads to an increased central aortic pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Treated or non-treated arterial hypertension
* History of cardiovascular disease
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
central aortic pressure | baseline
  effect of microgravity on central aortic blood pressure (measured in mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DP Denise, PhD, Principal Investigator — CHU CAEN
Locations (1):
- Caen CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No